CLINICAL TRIAL: NCT01791647
Title: Myo-inositol Versus Metformin: Effects of Six Months Treatment on Clinical, Endocrine and Metabolic Features in Obese Women With Polycystic Ovary Syndrome
Brief Title: Myo-inositol Versus Metformin in Obese Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Maurizio Guido, principal investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000102011
Record Dates: First submitted 2012-03-12; First posted 2013-02-15 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; myoinositol; metformin; glucose-insulinemic metabolism; menstrual pattern; insulin-lowering therapies
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Inositol

ARMS (2):
- myo-inositol (Active Comparator): 1500 mg/day myoinositol
  Interventions: Drug: myoinositol 1500 mg
- metformin (Active Comparator): 1500 mg/day of metformin
  Interventions: Drug: metformin 1500 mg

INTERVENTIONS:
Drug: metformin 1500 mg
  Arms: metformin
Drug: myoinositol 1500 mg
  Arms: myo-inositol

SUMMARY:
The aim of this study is to compare the effects of six months treatment of two insulin-lowering therapies on the clinical and endocrine-metabolic parameters in obese women affected by polycystic ovary syndrome. The study group includes 40 patients, randomly allocated to subgroup A (metformin 1500 mg/day) and subgroup B (myo-inositol 1500 mg/day). The investigations include menstrual pattern and hirsutism score evaluation, hormonal assays, oral glucose tolerance test, euglycemic hyperinsulinaemic clamp and lipid profile at baseline and after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with Polycystic Ovary Syndrome, diagnosed in accordance with Rotterdam Consensus Conference Criteria 2003;
* BMI>25 kg/m2;
* age 18-35 years.

Exclusion Criteria:

* pregnancy;
* significant liver or renal impairment;
* other hormonal dysfunction (hypothalamic, pituitary, thyroidal or adrenal causes for the clinical signs);
* neoplasms;
* unstable mental illness;
* diagnosis of diabetes mellitus or impaired glucose tolerance;
* use of drugs able to interfere with gluco-insulinaemic metabolism for at least three months prior to entering the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
number of cycles | six months

SECONDARY OUTCOMES:
effects of two therapies on glyco-insulinemic metabolism | six months
  Area under the curve insulin post oral glucose tolerance test (μUI/ML/180min), M value of euglycemic hyperinsulinaemic clamp(mg/kg/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy